CLINICAL TRIAL: NCT03582072
Title: Contacting GPs to Reduce Unnecessary Prescriptions of Antibiotics
Brief Title: CMO Letter to Reduce Unnecessary Antibiotic Prescribing March 2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CMO letter March 2018
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2018-04

CONDITIONS: Prescribing, Off-Label

STUDY DESIGN:
Intervention Model Description: 930 practices (this will be the number of datapoints), 478 in the intervention, 452 in the control; letter sent to individual GPS (4796 subjects, as below), 2340 in the intervention, 2456 in the control
  practices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- letter (Experimental): letter from the CMO: practice outside the top 20% of prescribers whose prescribing increased by > 4%, where GPs in the practice were sent a letter informing them their prescribing had increased
  Interventions: Behavioral: letter from the CMO
- control (No Intervention): practice outside of the top 20% of prescribers whose prescribing increase by >4%, GPs were not sent a letter

INTERVENTIONS:
Behavioral: letter from the CMO — informed GPs that: The great majority (80%) of practices in England reduced or stabilised their antibiotic prescribing rates in 2016/17. However, your practice is in the minority that have increased their prescribing by more than 4%.*
  Arms: letter

SUMMARY:
This trial aims to reduce unnecessary prescription of antibiotics by general practitioners (GPs) in England. Unnecessary prescriptions are defined as those that do not improve patient health outcomes. The intervention is to send GPs a letter from the Chief Medical Officer (CMO) that gives feedback on their practice's prescribing levels. Specifically, GPs in practices whose prescribing has increase by more than 4% over the past year will receive a letter stating that "The great majority (80%) of practices in England reduced or stabilised their antibiotic prescribing rates in 2016/17. However, your practice is in the minority that have increased their prescribing by more than 4%." The letter will also contain a leaflet to help GPs discuss self-care advice with patients and some advice to use delayed prescriptions. The investigators hypothesize that the antibiotic prescribing rate in will be lower for the treatment group compared to the control group, following the receipt of the letter.

DETAILED DESCRIPTION:
The investigators hypothesize that the antibiotic prescribing rate in will be lower for the treatment group compared to the control group; the statistical analysis will compare prescribing in March, April, and over the summer (treating May-September as a single data point).

ELIGIBILITY:
Inclusion Criteria:

* GP practices that increased the number of prescriptions in the financial year 2016/17, compared to the baseline of financial year 2015/16, by 4% or more

Exclusion Criteria:

* GP practices are excluded if their current level of prescription (doses per 1000 head of population) is classed as an outlier. The cut off for outliers is made at the 95th percentile of the distribution.
* Practices that have not been open since at least October 2013 will be excluded. This is because they will lack the historical data necessary to apply a control for seasonal effects to the main outcome variable.
* practices whose antibiotic prescribing rate is in the top 20% for their National Health Service (NHS) Local Area, controlling for relevant patient characteristics.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4796 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
antibiotic prescribing in March | 1 month
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
antibiotic prescribing in April | 2 months
  antibiotic prescribing weighted by STAR-PU
antibiotic prescribing May-September | 3-7 months
  antibiotic prescribing weighted by STAR-PU

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health England, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no individual participant data (IPD). The outcome measure is practice-level prescribing data, which is already publicly available.